CLINICAL TRIAL: NCT06307613
Title: A Phase 3, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Efgartigimod PH20 SC Administered by Prefilled Syringe in Adult Participants With Thyroid Eye Disease
Brief Title: A Study of Efgartigimod PH20 SC Given by Prefilled Syringe in Adults With Thyroid Eye Disease
Acronym: UplighTED
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2301; 2023-509197-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod arm (Experimental): Participants with active, moderate-to-severe TED receiving Efgartigimod PH20 SC (subcutaneously) via pre-filled syringe (PFS)
  Interventions: Combination Product: Efgartigimod PH20 SC
- Placebo arm (Placebo Comparator): Participants with active, moderate-to-severe TED receiving Placebo PH20 SC (subcutaneously) via pre-filled syringe (PFS)
  Interventions: Other: Placebo PH20 SC

INTERVENTIONS:
Combination Product: Efgartigimod PH20 SC — Subcutaneous efgartigimod PH20 SC given by prefilled syringe
  Arms: Efgartigimod arm
Other: Placebo PH20 SC — Subcutaneous placebo given by prefilled syringe
  Arms: Placebo arm

SUMMARY:
This study aims to evaluate the efficacy, safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of efgartigimod PH20 SC in participants with active, moderate-to-severe TED, compared with placebo PH20 SC.

After the screening period, eligible participants will be randomized in a 2:1 ratio to receive efgartigimod PH20 SC or placebo PH20 SC, respectively during the double-blinded treatment period (DBTP). At the end of the DBTP, participants may enter a follow-up observational period while off study drug. Some participants may also enter the open-label treatment period with efgartigimod PH20 SC. The study duration varies from approximately 60 to 110 weeks.

An alternative list of clinical sites open for recruitment could be found in the other UplighTED study record (https://www.clinicaltrials.gov/study/NCT06307626).

This study was terminated early on 15 December 2025 as the pre-defined interim analysis concluded that continuing the trials is unlikely to demonstrate the intended efficacy. This decision is not related to safety concerns, and the safety profile of efgartigimod remains unchanged. End-of-study and Safety-Follow-Up visits are ongoing for the participants of this trial.

ELIGIBILITY:
Inclusion Criteria:

* The participant is at least 18 years of age
* The participant is capable of providing signed informed consent and following with protocol requirements
* The investigator determines active, moderate-to-severe thyroid eye disease (TED) associated with autoimmune thyroid conditions (Graves' disease or Hashimoto's thyroiditis) for the most severely affected eye
* The participant has first onset of active TED symptoms within 12 months before screening
* The participant must have normal thyroid function with the baseline disease under control or have mild hypo or hyperthyroidism at screening. Every effort should be made to correct the mild hypo or hyperthyroidism promptly and to maintain the normal thyroid function for the full duration of the study
* The participant agrees to use birth control consistent with local regulations and the people of child-bearing potential must have a negative blood pregnancy test at screening and a negative urine pregnancy test before receiving the study drug

Exclusion Criteria:

* Optic neuropathy (damage to optic nerve), defined as new visual field defect (blind spot), relative afferent pupillary defect (pupils respond differently to light), or color defect secondary to optic nerve involvement within the 6 months before screening
* Corneal decompensation (swelling of the cornea) unresponsive to medical management
* Previous orbital irradiation or surgery for TED
* Use of some medications before screening (more information is found in the protocol)
* Known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of TED or puts the participant at undue risk
* History of malignancy, cancer, unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological findings of prostate cancer
* Clinically significant active infection that is not sufficiently resolved in the investigator's opinion or positive serum test at screening for active infection with any of the following: Hepatitis B virus (HBV), Hepatitis C virus (HCV), HIV
* Current participation in another interventional clinical study or previous participation in an efgartigimod clinical study and at least 1 dose of study drug received or has received at least 1 dose of commercially available efgartigimod
* Known hypersensitivity to study drug or one of its excipients (inactive ingredients)
* History of or current alcohol, drug, or medication abuse within 12 months before screening as assessed by the investigator
* Pregnant or lactating state or intention to become pregnant during the study
* Live or live-attenuated vaccine received <4 weeks before screening

The complete list of exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were proptosis responders | At week 24 of the Double-Blinded Treatment Period

SECONDARY OUTCOMES:
Change in proptosis measurement in the study eye from baseline | Up to week 24 of the Double-Blinded Treatment Period
Change in the total Graves' Orbitopathy Quality of Life (GO-QoL) score from baseline | Up to week 24 of the Double-Blinded Treatment Period
  Minimum value: 0 (most negative impact on Quality of Life); Maximum value: 100 (No impact on Quality of Life)
Percentage of participants with a resolution of diplopia (responders) | At week 24 of the Double-Blinded Treatment Period

CONTACTS AND LOCATIONS:
Locations (77):
- United States (16):
  - Thrive Health - Beverly Hills, Beverly Hills, California
  - UCI Health - Gavin Herbert Eye Institute, Irvine, California
  - University Of Southern California - Keck School Of Medicine, Los Angeles, California
  - Silkiss Eye Surgery, San Francisco, California
  - Advanced Research LLC, Coral Springs, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - University of South Florida (USF) Health - Morsani Center for Advanced Healthcare, Tampa, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - Wilmer Eye Institute, Baltimore, Maryland
  - University of Michigan, Ann Arbour, Michigan
  - Moyes Eye Center - Northland, Kansas City, Missouri
  - Quest Diagnostics - Mercy Smith Glynn Callaway, Springfield, Missouri
  - Duke University, Durham, North Carolina
  - Penn Medicine - Penn Presbyterian Medical Center - Scheie Eye Institute, Philadelphia, Pennsylvania
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Australia (4):
  - Centre for Eye Research Australia, Melbourne
  - The University of Western Australia - Lions Eye Institute (LEI), Nedlands
  - North Shore Private Hospital, St Leonards
  - Sydney Eye Hospital, Sydney
- CHU UVC Brugmann - Site Victor Horta, Brussels, Belgium
- Bulgaria (4):
  - Oxycom Medical Centre, Burgas
  - UMHAT Aleksandrovska - Diagnostic Consultative Center (DCC) Aleksandrova, Sofia
  - Medical Center Vereya EOOD - Vereya Medical Center (former Military Hospital), Stara Zagora
  - St. Petka Eye Hospital - Eye Clinic St. Petka Varna, Varna
- China (8):
  - Peking Union Medical College Hospital - Dongdan campus, Beijing
  - Shunde Hospital of Southern Medical University, Foshan
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Shanghai Ninth People's Hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Hospital of China Medical University, Shenyang
- Czechia (4):
  - Fakultni Nemocnice Olomouc - Ocni Klinika, Olomouc
  - OFTEX - Ocni klinika, Pardubice
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Axon Clinical s.r.o, Prague
- Estonia (2):
  - Dr Liina Viitas Endokrinoloog, Pärnu
  - Tartu Ulikooli Kliinikum, Tartu
- Germany (4):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Buergerhospital Frankfurt am Main, Frankfurt
  - Universitaetsklinikum der Ernst-Moritz-Arndt-Universitaet Greifswald, Greifswald
  - Universitaetsklinikum Muenster, Münster
- Greece (4):
  - General Hospital of Athens G Gennimatas, Athens
  - University General Hospital of Patras, Pátrai
  - A.LOUKAS General Hospital of Thessaloniki, Thessaloniki
  - Athens Medical Group - European Interbalkan Medical Center, Thessaloniki
- Hungary (5):
  - Budapest Retina Intezet, Budapest
  - Vadnay Szemeszet es Latszereszet, Eger
  - Ganglion Orvosi Kozpont, Pécs
  - Pecsi Tudomanyegyetem (PTE) Altalanos Orvostudomanyi Kar (AOK) University of Pecs Medical School, Pécs
  - Markusovszky Teaching Hospital, Szombathely
- Italy (7):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - Fondazione Irccs Ca' Granda Ospedale Maggioe Policlinico Di Milano, Milan
  - ASST Santi Paolo e Carlo - Ospedale San Paolo, Milan
  - Azienda Ospedaliera Universitaria (AOU) Federico II, Naples
  - Santa Chiara Hospital, Pisa
  - ASST Sete Laghi - Ospedale di Circolo e Fondazione Macchi di Varese, Varese
- Romania (4):
  - Centrul Medical Sana, Bucharest
  - Institutul National de Endocrinologie C.I.Parhon, Bucharest
  - Spitalul Universitar De Urgenta Militar Central Dr. Carol Davila, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Spiridon, Iași
- National University Hospital, Singapore, Singapore
- Spain (4):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bang Phlat
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- United Kingdom (5):
  - Bradford Royal Infirmary - Bradford Teaching Hospitals NHS Foundation, Bradford
  - Cardiff and Vale University Health Board - University Hospital of wales (UHW), Cardiff
  - Frimley Health NHS Foundation Trust - Frimley Park Hospital, Frimley
  - St Thomas' Hospital - Guy's & St Thomas' NHS Foundation Trust, London
  - Royal Victoria Infirmary - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle